CLINICAL TRIAL: NCT00183092
Title: Novel Therapeutics For Prion Diseases: A Randomized, Double-blinded, Placebo-controlled Study of the Efficacy of Quinacrine in the Treatment of Sporadic Creutzfeldt-Jakob Disease
Brief Title: CJD (Creutzfeldt-Jakob Disease) Quinacrine Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IA0083; P01AG021601 (NIH)
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Results first posted 2014-05-29 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Creutzfeldt-Jakob Disease
Keywords: dementia; spongiform encephalopathy; nervous system disorder; acridine; prion; neuropharmacologic agent
MeSH Terms: conditions — Creutzfeldt-Jakob Syndrome; Dementia; Prion Diseases; Nervous System Diseases; Insomnia, Fatal Familial | interventions — Quinacrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- quinacrine (Experimental)
  Interventions: Drug: Quinacrine
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quinacrine — 100mg by mouth three times a day
  Other Names: Atabrine
  Arms: quinacrine
Drug: Placebo — 100mg by mouth three times a day
  Arms: placebo

SUMMARY:
The purpose of this clinical trial is to determine the effectiveness of the medication quinacrine on survival in sporadic Creutzfeldt-Jakob disease (sCJD).

DETAILED DESCRIPTION:
Creutzfeldt-Jakob disease (CJD)is a rapidly progressive, invariably fatal and untreatable neurodegenerative disease with a mean duration of about eight months. Beyond the debilitating cognitive and motor deficits that accompany CJD, the difficulty in treating behavioral and mood disturbances and the rapidity of its course compound its tragedy. Recent results from experiments show that, at physiological concentrations, the anti-malarial drug quinacrine permanently clears abnormal prion proteins from cell culture. The demonstrated efficacy of quinacrine in cell culture, its relative safety and well known side-effects in the clinical setting, and the universal fatality of CJD justify quinacrine as an immediate candidate for the treatment of CJD.

The purpose of this clinical trial is to determine the efficacy of the medication quinacrine on survival in sporadic CJD (sCJD). This will be accomplished by bringing approximately 60 patients with probable or definite sCJD over approximately three years to UCSF for evaluation and initiation of a randomized, double-blinded, placebo-controlled (delayed treatment start) treatment study of quinacrine. Each patient will have a 50:50 chance of being placed on quinacrine or placebo upon study enrollment; however, all patients will be offered quinacrine after two months. Prior to study enrollment, patients will have a comprehensive clinical assessment to confirm the diagnosis of sCJD. Participants will come to UCSF for initial evaluation, potential study enrollment and, if possible, return to UCSF for follow-up at two and twelve months. Patients will receive telephone follow-up (every 2 weeks for the first two months and monthly thereafter) and local blood and testing to monitor for possible medication toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable or definite sCJD: Definite--biopsy confirmed sCJD; Probable--a progressive dementia with either a typical EEG or a typical MRI consistent with sCJD, and at least two of the following clinical features: myoclonus, pyramidal or extrapyramidal signs, visual symptoms, cerebellar signs, akinetic mutism, other focal higher cortical neurologic signs (e.g. neglect, apraxia, aphasia)
* 18 years of age or older
* Able to swallow
* Able to follow simple one-step commands
* Have had a brain MRI within 6 months and an EEG within 3 months ruling out other etiologies such as masses, strokes, or non-convulsive status epilepticus
* Consent to autopsy in the event of their death during or after the study

Exclusion Criteria:

* History of other significant or life-threatening disease, including: cancer; end-stage liver or renal disease; severe heart disease
* History of other disease requiring regular supportive care
* Liver disease
* Active alcoholism
* Bone marrow suppression
* Severe hypotension
* Severe psoriasis
* Poorly controlled diabetes
* Women who are pregnant or breast-feeding
* Men, or women of childbearing age, not practicing reliable contraception
* Serious allergies to quinacrine or other acridines
* Current or recent use of quinacrine (within 6 months)
* < 18 years of age
* Any other contraindication to taking quinacrine
* Genetic form of prion disease is identified prior to study enrollment
* Current use of anti-arrhythmics (at discretion of investigator)
* G6PD (Glucose 6-Phosphate Dehydrogenase) deficiency (at discretion of investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2005-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Geschwind, MD, PhD, Principal Investigator — UCSF Memory & Aging Center, University of California, San Francisco; Bruce L. Miller, MD, Principal Investigator — UCSF Memory & Aging Center, University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Prusiner SB. Prions. Proc Natl Acad Sci U S A. 1998 Nov 10;95(23):13363-83. doi: 10.1073/pnas.95.23.13363. PMID 9811807
- [Background] Korth C, May BC, Cohen FE, Prusiner SB. Acridine and phenothiazine derivatives as pharmacotherapeutics for prion disease. Proc Natl Acad Sci U S A. 2001 Aug 14;98(17):9836-41. doi: 10.1073/pnas.161274798. PMID 11504948
- [Background] Scoazec JY, Krolak-Salmon P, Casez O, Besson G, Thobois S, Kopp N, Perret-Liaudet A, Streichenberger N. Quinacrine-induced cytolytic hepatitis in sporadic Creutzfeldt-Jakob disease. Ann Neurol. 2003 Apr;53(4):546-7. doi: 10.1002/ana.10530. No abstract available. PMID 12666126
- [Background] Wallace DJ. Is there a role for quinacrine (Atabrine) in the new millennium? Lupus. 2000;9(2):81-2. doi: 10.1191/096120300678828163. No abstract available. PMID 10787002
- [Background] Engel GL. Quinacrine effects on the central nervous system. JAMA. 1966 Aug 8;197(6):515. No abstract available. PMID 5952734
- [Derived] Geschwind MD, Kuo AL, Wong KS, Haman A, Devereux G, Raudabaugh BJ, Johnson DY, Torres-Chae CC, Finley R, Garcia P, Thai JN, Cheng HQ, Neuhaus JM, Forner SA, Duncan JL, Possin KL, Dearmond SJ, Prusiner SB, Miller BL. Quinacrine treatment trial for sporadic Creutzfeldt-Jakob disease. Neurology. 2013 Dec 3;81(23):2015-23. doi: 10.1212/WNL.0b013e3182a9f3b4. Epub 2013 Oct 11. PMID 24122181
- See also: UCSF Memory & Aging Center — http://memory.ucsf.edu
- See also: UCSF Institute for Neurodegenerative Diseases — http://ind.universityofcalifornia.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in April 2005 and ended in January 2009. Subjects came from across the USA, as well as Canada, with a plurality from California, and enrolled at one U.S. clinical site (University of California, San Francisco).
Pre-assignment Details: 425 patients referred; 69 subjects consented/enrolled; 54 subjects eligible/randomized; 3 randomized subjects identified as carriers of PrP (prion protein) gene mutations as determined by analysis of sequence variability of the bovine prion protein gene (PRNP) and excluded from analyses.
Groups:
- Quinacrine: Double Blind Period: 100mg Quinacrine by mouth three times a day. Open Label Period: Choice of study drug or open-label Quinacrine 100mg by mouth three times a day.
- Placebo: Double Blind Period: 100mg Placebo by mouth three times a day. Open Label Period: Choice of study drug or Quinacrine 100mg by mouth three times a day.
- Study Drug (Quinacrine) During Open-Label Period: Participants received Quinacrine during Double-Blind period and opted to continue study drug during Open-Label period
- Study Drug (Placebo) During Open-Label Period: Participants received Placebo during Double-Blind period and opted to continue study drug during Open-Label period
Period: Double-blind (Baseline - Month 2)
Arm/Group | Quinacrine | Placebo | Study Drug (Quinacrine) During Open-Label Period | Study Drug (Placebo) During Open-Label Period
Started | 23 | 28 | 0 | 0
Alive at Month 2 | 13 | 19 | 0 | 0
Came in for Month 2 Visit | 10 | 16 | 0 | 0
Completed | 11 | 16 | 0 | 0
Not Completed | 12 | 12 | 0 | 0
Period: Open-label Period (Month 2 Until Death)
Arm/Group | Quinacrine | Placebo | Study Drug (Quinacrine) During Open-Label Period | Study Drug (Placebo) During Open-Label Period
Started | 10 (Participants initially assigned to Quinacrine opted to begin open-label Quinacrine at Month 2) | 14 (Participants initially assigned to Placebo opted to begin open-label Quinacrine at Month 2) | 1 (Participants assigned to Quinacrine opted to continue assigned drug during open-label period) | 1 (Participants assigned to Placebo opted to continue assigned drug during open-label period)
Completed | 0 | 0 | 0 | 0
Not Completed | 10 | 14 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo : 100mg by mouth three times a day
- Quinacrine: Quinacrine : 100mg by mouth three times a day
- Total: Total of all reporting groups
Arm/Group | Placebo | Quinacrine | Total
Number analyzed (Participants) | 28 | 23 | 51
Age, Continuous [Mean (Full Range); unit: years] | 64.4 (10.9) [38 to 82] | 60.5 (8.0) [40 to 75] | 62.5 [38 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 19 | 12 | 31
Region of Enrollment [Number; unit: participants]
  United States | 28 | 23 | 51

OUTCOME MEASURES:

1. Primary Outcome: Primary Survival
Description: Participants alive after 2 months on study treatment
Time Frame: Randomization to Month-2
Measure: Number; unit: participants
Arm/Group | Placebo | Quinacrine
Number analyzed (Participants) | 28 | 23
participants | 19 | 13
Statistical Analysis 1: Comparison: Placebo vs Quinacrine; Test type: Superiority or Other; p = 0.43, Regression, Cox; Cox Proportional Hazard = 1.43, 95% CI 2-sided [0.58 to 3.53]

2. Secondary Outcome: Change in Mini-Mental State Examination (MMSE) After 2 Months
Description: The mini-mental state examination (MMSE) is a brief 30-point questionnaire that is used to screen for cognitive impairment. In about 10 minutes it samples functions including arithmetic, memory and orientation. A score greater than or equal to 25 points (out of 30) indicates a normal cognition. Lower scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-24 points) cognitive impairment. Low to very low scores correlate closely with the presence of dementia, although other mental disorders can also lead to abnormal findings on MMSE testing.
Time Frame: Baseline to Month-2
Population: Subjects still alive, who attended the month-2 visit and were willing and able to tolerate cognitive testing. 1 subject in each arm did attend the 2-month visit but did not cooperate fully with the MMSE, which was therefore not scored.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Placebo | Quinacrine
Number analyzed (Participants) | 15 | 9
units on a scale | -6.9 [-18 to 4] | -3.9 [-10 to 1]
Statistical Analysis 1: Comparison: Placebo vs Quinacrine; The difference between change scores, adjusted for Month-0 performance. Positive adjusted differences indicate greater adjusted change (worsening) in the placebo group; negative indicate greater adjusted changed (worsening) in the quinacrine group; Test type: Superiority or Other; p = .54, ANCOVA — Threshold for statistical significance = 0.05. One subject in the placebo group was administered only 25 items on the MMSE due to visual impairment, and this subject's score was scaled based on percentage correct; Mean Difference (Net) = 1.5

3. Secondary Outcome: Barthel Score Change After 2 Months
Description: An ordinal scale used to measure performance in activities of daily living. Scores range from 0 (worst, fully dependent) to 100 (best, independent); higher score associated with a greater likelihood of being able to live at home with a degree of independence following discharge from hospital. 10 individual items are scored and summed to derive the overall Barthel index score. Each item may be scored 0, 5, 10 or 15; not all items use the full range of 4 possible values. The amount of time and physical assistance required to perform each item are considered in scoring each item. For subjects unable to return for month-2 visit, Barthel Index was performed via telephone.
Time Frame: baseline, 2 months
Population: One surviving subject in the quinacrine arm did not attend the 2-month visit and was lost-to-followup; for a second surviving subject in the quinacrine arm, the Barthel Index was inadvertently not performed at the 2-month visit.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Placebo | Quinacrine
Number analyzed (Participants) | 19 | 11
units on a scale | -23.2 [-85 to 70] | -13.2 [-65 to 5]
Statistical Analysis 1: Comparison: Placebo vs Quinacrine; The difference between scores, adjusted for Month-0 performance; Test type: Superiority or Other; p = .36, Quade's rank analysis of covariance — significance threshold p=0.05; Mean Difference (Net) = 7.9

4. Secondary Outcome: Change in Clinical Dementia Rating Scale Sum of Boxes (CDRS-SB) After 2 Months
Description: Clinical Dementia Rating Scale Sum of Boxes (CDRS-SB). The CDR is obtained through semistructured interviews of patients and informants, and cognitive functioning is rated in 6 domains of functioning: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain is rated on a 5-point scale of functioning: 0, no impairment; 0.5, questionable impairment; 1, mild impairment; 2, moderate impairment; and 3, severe impairment (personal care is scored on a 4-point scale without a 0.5 rating available). The global CDR score is computed via an algorithm. The CDR-SB score is obtained by summing each of the domain box scores, with scores ranging from 0 to 18. A higher value and/or positive change is worse. For subjects unable to return for month-2 visit, CDRS-SB was performed via telephone.
Time Frame: Baseline, 2 months
Population: For subjects still alive at month 2 and assessed at the 2-month visit or via telephone
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Placebo | Quinacrine
Number analyzed (Participants) | 19 | 12
units on a scale | 3.2 [-1 to 8] | 0.3 [-1 to 2]
Statistical Analysis 1: Comparison: Placebo vs Quinacrine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = .01, Quade's rank analysis of covariance — Significance threshold p<0.05; Mean Difference (Net) = 2.8

5. Secondary Outcome: Change in Rankin Score After 2 Months
Description: The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead. For subjects unable to return for the 2-month visit, Rankin score was assessed via telephone.
Time Frame: Baseline, 2 months
Population: For subjects still alive at month 2 and assessed at the 2-month visit or via telephone
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Placebo | Quinacrine
Number analyzed (Participants) | 19 | 12
units on a scale | 0.8 [0 to 2] | 0.3 [-1 to 2]
Statistical Analysis 1: Comparison: Placebo vs Quinacrine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.03, Quade's rank analysis of covariance — Threshold for significance p<0.05; Mean Difference (Net) = 0.5

6. Secondary Outcome: ADAS-Cog Change After 2 Months Among Survivors
Description: ADAS-cog measures cognitive performance by combining ratings of 11 components (word recall, word recognition, constructional praxis, orientation, naming objects and fingers, commands, ideational praxis, remembering instruction, spoken language, word finding, comprehension) representing six areas of cognition: memory; language; orientation to time, place and person; construction of simple designs and planning; and performing simple behaviors in pursuit of a basic, predefined goal. Seven components are scored as the 'number incorrect'. For example, in the commands component, the number of five commands performed incorrectly (range: 0-5). Four components are scored from 0 (no limitations) to 5 (max limitations) as the examiner's perception of remembering instructions, spoken language ability, word finding and comprehension. Component scores are summed into a total ADAS-cog score ranging from 0-75, with low scores indicating better cognitive performance.
Time Frame: Baseline, 2 months
Population: Subjects still alive and able to tolerate cognitive testing at Month 2 visit.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Placebo | Quinacrine
Number analyzed (Participants) | 9 | 4
units on a scale | 13.0 [0 to 23] | 12.6 [-2 to 37]
Statistical Analysis 1: Comparison: Placebo vs Quinacrine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.92, ANCOVA — Significance threshold p<0.05; Mean Difference (Net) = -0.7

7. Secondary Outcome: Change in Phonemic Fluency (Words Beginning With Letter "D")
Description: Verbal fluency tests are a kind of psychological test in which participants have to say as many words as possible from a category in 60 seconds. This category (words beginning with letter "D") is phonemic. Higher scores indicate better cognition.
Time Frame: Baseline, 2 months
Population: Subject still alive and able to tolerate cognitive testing at month 2 visit
Measure: Mean (Full Range); unit: number of words generated
Arm/Group | Placebo | Quinacrine
Number analyzed (Participants) | 9 | 5
number of words generated | -2.4 [-8 to 1] | -2.2 [-5 to 0]
Statistical Analysis 1: Comparison: Placebo vs Quinacrine; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.71, ANCOVA — Significance threshold p<0.05; Mean Difference (Net) = 0.4

8. Secondary Outcome: Change in Semantic Verbal Fluency (Naming Animals)
Description: Verbal fluency tests are a kind of psychological test in which participants have to say as many words as possible from a category in 60 seconds. This category (naming animals) is semantic. Higher scores indicate better cognition.
Time Frame: Baseline, 2 months
Population: Subjects still alive and able to tolerate cognitive testing at month 2 visit.
Measure: Mean (Full Range); unit: number of words generated
Arm/Group | Placebo | Quinacrine
Number analyzed (Participants) | 9 | 5
number of words generated | -3.2 [-9 to 2] | -2.2 [-9 to 5]
Statistical Analysis 1: Comparison: Placebo vs Quinacrine; The difference between change scores, adjusted for Month-0 performance. Positive adjusted differences indicate greater adjusted change (worsening) in the placebo group; negative indicate greater adjusted change (worsening) in the quinacrine group; Test type: Superiority or Other; p = 0.70, ANCOVA — Significance threshold p<0.05; Mean Difference (Net) = 0.8

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Placebo Random Assignment: Placebo : 100mg by mouth three times a day, Baseline-Month 2 = random assignment (n=28), Month 2+ = optional continuation of assigned drug (n=1).
- Quinacrine Random Assignment: Quinacrine: 100mg by mouth three times a day. Baseline-Month 2 = random assignment (n=23), Month 2+ = optional continuation of assigned drug (n=1).
- Quinacrine Open-label: Quinacrine: Month 2 until death = optional open-label Quinacrine 100mg by mouth three times a day
Arm/Group | Placebo Random Assignment | Quinacrine Random Assignment | Quinacrine Open-label
Serious Adverse Events (participants affected / at risk) | 14/28 | 13/23 | 14/24
Other Adverse Events (participants affected / at risk) | 9/28 | 9/23 | 16/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Random Assignment (N=28) | Quinacrine Random Assignment (N=23) | Quinacrine Open-label (N=24)
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhage (Nervous system disorders) | 1 | 0 | 1 — Hemorrhagic brain bleed found on autopsy
Death (General disorders) | 11 | 10 | 8
Seizure (Nervous system disorders) | 0 | 1 | 0
Unclassified shaking (General disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 — Present prior to randomization
Elevated renal function labs (Renal and urinary disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Post-LP infection (Injury, poisoning and procedural complications) | 2 | 0 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 1
Post-LP headache (Injury, poisoning and procedural complications) | 2 | 0 | 0
Post-LP Dizziness (Injury, poisoning and procedural complications) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Random Assignment (N=28) | Quinacrine Random Assignment (N=23) | Quinacrine Open-label (N=24)
Abdominal abscess (Gastrointestinal disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 2 | 2
Elevated Liver Function Tests (Hepatobiliary disorders) | 0 | 3 | 12
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 5
Urinary Tract Infection (Infections and infestations) | 3 | 1 | 1
Potential thrombi (Blood and lymphatic system disorders) | 1 | 0 | 1 — Present prior to randomization
Post-LP complications (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hallucination (Psychiatric disorders) | 2 | 0 | 0
Pulmonary embolism (Blood and lymphatic system disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Elevated creatine kinase (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (General disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 5
Vomiting (Gastrointestinal disorders) | 1 | 1 | 5
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Fever (General disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes